CLINICAL TRIAL: NCT01087658
Title: A Multicentre, Randomized, Open-label, Phase III Study Comparing the Efficacy of Oral Glutamine and Calcium-magnesium With Calcium-magnesium Alone in the Prevention of Oxaliplatin-induced Neurotoxicity in Patients With Colorectal Cancer Treated With Oxaliplatin in Adjuvant or 1st Line Metastatic Settings.
Brief Title: Oral Glutamine in the Prevention of Oxaliplatin-induced Neurotoxicity
Acronym: GLUTOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXALI_L_03768; U1111-1116-9494 (Other: UTN)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Glutamine; Calcium; Magnesium

ARMS (2):
- Glutamine and calcium magnesium (Experimental): Glutamine 10g p.o. 3-times a day beginning at day -2 for 7 consecutive days during each chemotherapy cycle. 1g of calcium and 1g of magnesium i.v. over 30 minutes just before the chemotherapy and repeated at the same dose after the completion of the oxaliplatine infusion.
  All patients will receive an oxaliplatin based chemotherapy with XELOX, FOLFOX-4 or mFOLFOX-6.
  Interventions: Drug: Glutamine; Drug: Calcium and Magnesium
- Calcium magnesium (Active Comparator): 1g of calcium and 1g of magnesium i.v. over 30 minutes just before the chemotherapy and repeated at the same dose after the completion of the oxaliplatine infusion.
  All patients will receive an oxaliplatin based chemotherapy with XELOX, FOLFOX-4 or mFOLFOX-6.
  Interventions: Drug: Calcium and Magnesium

INTERVENTIONS:
Drug: Glutamine — Per os
  Arms: Glutamine and calcium magnesium
Drug: Calcium and Magnesium — Intravenous

SUMMARY:
Primary Objective:

To assess the benefit of glutamine when added to calcium-magnesium on the occurrence of grade 2, 3 and 4 peripheral sensory neuropathy (PSN) related to oxaliplatin with the National Cancer Institute-Common Terminology Criteria for Adverse Event (NCI-CTCAE) scale taking into account the time from start of oxaliplatin at which the first event occurred.

Secondary Objective:

To determine cumulative dose of oxaliplatin and time when the first occurrence of grade 2, 3 or 4 PSN.

To determine the incidence of dose-reductions, dose-delays and discontinuations of oxaliplatin due to PSN grade 3 or 4.

To assess effects of glutamine when added to calcium-magnesium on patients-reported outcomes using the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity 12 items questionnaire (FACT/GOG NTX-12) subscale.

To evaluate the incidence of diarrhea. To determine Progression Free Survival (PFS) in metastatic patients.

ELIGIBILITY:
Inclusion criteria:

1. Histologically- or cytologically- proven adenocarcinoma of the colon or rectum.
2. Disease either in adjuvant or 1st line metastatic setting.
3. Eastern Cooperation Oncology Group (ECOG) performance status inferior or equal to 2.
4. At least 4 weeks following any major surgical procedure(s) and recovery from any surgical sequelae.
5. Electrocardiogram (ECG) with no acute or recent changes within limit of normal range, and not presenting abnormalities contraindicating the proposed chemotherapy.
6. Adequate liver and kidney function:

   * Total bilirubin inferior to 1.5 ULN
   * Serum creatinine inferior to 150 umol/L
   * Creatinine clearance (ClCr) superior to 45 mL/min
   * ALT/AST inferior to 3 ULN
   * Alkaline phosphatase inferior or equal to 2 ULN, unless liver metastases are present and documented at baseline by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) scans (inferior or equal to 3,5 ULN in that case).
7. Adequate hematological function:

   * Neutrophils superior or equal to 1.5 x 109/L
   * Platelet count superior or equal to 100 x 109/L
   * Hemoglobin superior to 9 g/dL

Exclusion criteria:

1. Any condition or past medical history that contra-indicates treatment with oxaliplatin, 5-fluorouracil (5-FU), leucovorin (LV) or capecitabine as reported in the approved labeling information.
2. Previous oxaliplatin-based chemotherapy.
3. Previous or current diagnosis of PSN.
4. Concomitant treatments with drugs/ingredients reported to have a potential activity in preventing PSN: carbamazepine, amitriptyline, gabapentin, phenytoin, glutathione, alpha-lipoic acid, celecoxib, amifostine, venlafaxine, vitamin B1 (thiamine), B6 (pyridoxine).
5. History of known allergy to oxaliplatin or other platinum agents, 5-FU, LV or capecitabine.
6. History of known allergy to glutamine or to calcium-magnesium.
7. Participation in another clinical trial with any investigational drug within 30 days prior to study screening.
8. Uncontrolled intercurrent illness: e.g. high blood pressure, unstable angina, symptomatic congestive heart failure (New York Heart Association Classification III or IV),
9. Serious cardiac arrhythmia, diabetes, or active infection.
10. Concurrent active cancer originating from a primary site other than colon or rectum.
11. Presence of any symptom suggesting brain metastasis.
12. Patients who are pregnant or breast-feeding
13. Patients (males and females) with reproductive potential not implementing accepted and effective method of contraception
14. For patient who will receive Bevacizumab: Bevacizumab is contraindicated in patients with known hypersensitivity to any components of the product to Chinese hamster ovary cell product or other recombinant human or humanized antibodies

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Occurence of peripheral sensory neuropathy (PSN) grade 2, 3 and 4 assessed by the National Cancer Institute Common Terminology Criteria for Adverse Event (NCI-CTCAE) | Every cycle i.e. 2 or 3 weeks according to the treatment arm

SECONDARY OUTCOMES:
Cumulative dose of oxaliplatin and time of onset when the first PSN grade 2, 3 or 4 occurs | Every cycle i.e. 2 or 3 weeks according to the treatment arm
Dose-reduction, dose-delay and discontinuation of oxaliplatin due to PSN grade 3 or 4 | Every cycle i.e. 2 or 3 weeks according to the treatment arm
Patient self-reported neurotoxicity scale for chronic peripheral neuropathy | Every cycle i.e. 2 or 3 weeks according to the treatment arm
Progression Free Survival / PFS (for metastatic patients) | Every cycle i.e. 2 or 3 weeks according to the treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (14):
- Canada (14):
  - Investigational Site Number 0001, Greenfield Park
  - Investigational Site Number 124-005, Laval
  - Investigational Site Number 124-007, London
  - Investigational Site Number 124-014, Moncton
  - Investigational Site Number 124-006, Montreal
  - Investigational Site Number 124-004, Montreal
  - Investigational Site Number 124010, Montreal
  - Investigational Site Number 124-011, Montreal
  - Investigational Site Number 124-015, Oshawa
  - Investigational Site Number 124-012, Ottawa
  - Investigational Site Number 124-003, Québec
  - Investigational Site Number 124-017, Rimouski
  - Investigational Site Number 124-002, Toronto
  - Investigational Site Number 124-016, Winnipeg